CLINICAL TRIAL: NCT05184010
Title: Arthroscopic Treatment With and Without Ulnar Nerve Release for Elbow Osteoarthritis --a Prospective Randomized Controlled Trial
Brief Title: Arthroscopic Treatment With Ulnar Nerve Release for Elbow Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Lu
Record Dates: First submitted 2021-11-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Primary Osteoarthritis, Elbow; Ulnar Nerve Release

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthroscopic release with ulnar nerve mini open release (Experimental)
  Interventions: Device: ulnar nerve mini open release
- arthroscopic release alone without ulnar nerve mini open release (Placebo Comparator)
  Interventions: Device: without ulnar nerve mini open release

INTERVENTIONS:
Device: ulnar nerve mini open release — the ulnar nerve mini open release was performed before arthroscopic release for elbow
  Arms: arthroscopic release with ulnar nerve mini open release
Device: without ulnar nerve mini open release — arthroscopic release for elbow stiffness alone without ulnar nerve mini open release
  Arms: arthroscopic release alone without ulnar nerve mini open release

SUMMARY:
This study is a prospective randomized controlled study of arthroscopic release for primary osteoarthritis of the elbow with stiffness with or without ulnar nerve release. The patients with primary osteoarthritis of the elbow with stiffness, which ulnar neuropathy proven by electromyography without clinical symptoms, were randomly divided into groups before the operation. Before the arthroscopic operation was began, the procedure of ulnar nerve release was performed according to the group(release group or unrelease group). In different time periods postoperatively, the quantitative and qualitative indicators including pain, functional score, muscle strength, etc. were compared between groups at the same time period to evaluate the difference in the effect of arthroscopic treatment combined with ulnar nerve release.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Primary osteoarthritis of the elbow with stiffness. Osteoarthritis was confirmed on CT-arthrography, by cartilage damage, osteophytes or local or global joint impingement.
3. Ulnar neuropathy proven by electromyography without clinical symptoms
4. Failure at least 6 months of conservative treatment
5. Availability of medical information for >2 years of follow-up

Exclusion Criteria:

1. Severe skin contracture or wound problem that could affect the neurovascular structures or require flap surgery.
2. Revision surgery
3. Ulnar nerve pathology results in clinical symptom such as motion and feeling deficiency
4. Other indication for elbow arthroscopy: synovial or inflammatory rheumatoid pathology, osteochondritis dissecan, acute infection, tumor or pure capsular stiffness.
5. Inadequate or loss of follow-up
6. elbow instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
DASH | baseline-2 years postoperatively
  A score used to evaluated the elbow function,range of 0-100, 100 means worst outcome

SECONDARY OUTCOMES:
ROM(F-E and rotation) | baseline-2 years postoperatively
  the motion of the elbow
Strength | baseline-2 years postoperatively
  the strength test contain flex and extend the elbow, made a comparison with contralateral elbow.
MEPS | baseline-2 years postoperatively
  A score used to evaluated the elbow function

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No